CLINICAL TRIAL: NCT04610034
Title: "Resilient Caregivers" - A Randomized Controlled Trial of a Resilience-based Intervention for Distressed Partner Caregivers of Cancer Patients
Brief Title: "Resilient Caregivers" - A Resilience-based Intervention for Distressed Partner Cancer Caregivers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danish Cancer Society (Other)
Collaborators: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Pernille Bidstrup, Principle investigator, Danish Cancer Society
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Resilient Caregivers
Record Dates: First submitted 2020-09-27; First posted 2020-10-30 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Distress, Emotional
Keywords: Cancer caregivers; Distress; Anxiety; Resilience; Coping
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Resilient Caregivers" (Experimental): Intervention program
  Interventions: Behavioral: "Resilient Caregivers"
- Control group (Other): Care as usual
  Interventions: Other: Care as usual

INTERVENTIONS:
Behavioral: "Resilient Caregivers" — "Resilient Caregivers" is a 7-session group program developed for partner caregivers of patients with cancer (6 weekly sessions and 1 booster session). Each session takes place in groups of approximately 8 participants and lasts for two-and-a-half hours. Sessions 1 to 3 focuses on the caregiver and introduces the resilience components of coping strategies, meta-reflective skill and clarification of values. Sessions 4 and 5 focuses on these components in the relationship between the caregiver and the cancer patient and social support networks respectively, while Session 6 focuses on resilience in relation to self-care and care for the partner. A booster session will be scheduled one month after the end of Session 6 in order to follow-up on the intervention and allow participants to reflect on the benefits and challenges of the program.
  Arms: "Resilient Caregivers"
Other: Care as usual — The control arm will receive usual care, which implies no systematic support.
  Arms: Control group

SUMMARY:
The objective of this study is to develop and test the effectiveness of a resilience-based intervention for distressed partner caregivers of cancer patients in reducing symptoms of anxiety, depression and distress, while improving quality of life and resilience (meta-reflective skill, values clarification and coping strategies).

DETAILED DESCRIPTION:
Informal caregivers of cancer patients often experience significant psychological distress, which may even exceed that of the patient's. Partners or spouses are typically the most important caregiver and emotional support person for the cancer patient, but there is a lack of psychological interventions that specifically target caregiving partners. "Resilient Caregivers" is a novel 7-session group-based program aimed specifically at improving the participant's ability to cope with the stresses of being a partner to a cancer patient. In this randomized trial, the investigators aim to assess the potential efficacy of this program in improving the caregiver's resilience and quality of life, as well as reducing symptoms of anxiety, depression and distress. Outcomes will be assessed at baseline and at 3, 6 and 12-months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Partner/Spouse to a patient diagnosed with Stage I-III cancer and receiving cancer treatment at Herlev Hospital
* Patient performance status 1 or 2
* Distress Thermometer score > 4
* Able to speak and understand Danish
* Has given written informed consent to participate in the study

Exclusion Criteria:

* Being a cancer patient
* Has untreated psychopathology or physical impairment that may prevent attendance and participation in the study
* Active substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-03-19 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change in symptoms of anxiety | Baseline, 3 months, 6 months and 12 months follow-up
  Measured by Generalized Anxiety Disorder-7 (GAD-7); range 0-21; higher scores = more symptoms

SECONDARY OUTCOMES:
Change in psychological distress | Baseline, 3 months, 6 months and 12 months follow-up
  Measured by the Distress Thermometer; range 0-10; higher scores = higher distress
Change in symptoms of depression | Baseline, 3 months, 6 months and 12 months follow-up
  Measured by Patient Health Questionnaire-9 (PHQ-9); range 0-27; higher scores = more symptoms
Change in resilience | Baseline, 3 months, 6 months and 12 months follow-up
  Measured by Connor-Davidson Resilience Scale (CD-RISC-10); range 0-40; higher scores = greater resilience
Change in perceived stress | Baseline, 3 months, 6 months and 12 months follow-up
  Measured by Perceived Stress Scale (PSS-10); range 0-40; higher scores = higher perceived stress
Change in rumination/worry and coping | Baseline, 3 months, 6 months and 12 months follow-up
  Measured by Cognitive Attentional Syndrome Scale (CAS-1); range 0-100; higher scores = worse rumination/worry and coping
Change in quality of life | Baseline, 3 months, 6 months and 12 months follow-up
  Measured by World Health Organization-5 Well-being Index (WHO-5); range 0-25; higher scores = better quality of life
Change in valued living | Baseline, 3 months, 6 months and 12 months follow-up
  Measured by the "Obstruction subscale" from the Valuing Questionnaire (VQ); range 0-30; higher scores = more interference with living consistently with one's values
Change in sleep quality | Baseline, after completion of intervention (approximately 3 months from inclusion), 6 months and 12 months follow-up
  Measured by the Pittsburg Sleep Quality Index (PSQI); range 0-21; higher scores = worse sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Pernille Envold Bidstrup, Principal Investigator — Danish Cancer Society Research Center
Locations (1):
- Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Genter P, Hoeg BL, Hamre CJ, Andersen EAW, Dalton SO, Ribers B, Bidstrup PE. Protocol for 'Resilient Caregivers': a randomised trial of a resilience-based intervention for psychologically distressed partner caregivers of patients with cancer. BMJ Open. 2021 Nov 12;11(11):e048327. doi: 10.1136/bmjopen-2020-048327. PMID 34772747